CLINICAL TRIAL: NCT02329873
Title: Efficacy of the Respiratory Rehabilitation Exercise Training Package in Hospitalized Elderly Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease: Randomized Control Trial
Brief Title: Respiratory Rehabilitation Exercises in Older Adults With Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chest Hospital, Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Principal Investigator, Lin-Yu Liao, Head Nurse, Chest Hospital, Ministry of Health and Welfare, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ER-100-202
Record Dates: First submitted 2014-12-15; First posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Acute exacerbation of chronic obstructive pulmonary disease; Older adults; Respiratory rehabilitation exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Respiratory rehabilitation exercise training 2 times/day, 10-30 minutes per session for 4 days.
  Interventions: Behavioral: Respiratory rehabilitation exercise training
- Control group (No Intervention): Control group received usual care and health education.

INTERVENTIONS:
Behavioral: Respiratory rehabilitation exercise training — The respiratory rehabilitation exercise training package was conducted twice a day and 10-30 minutes per session for 4 days: (a) disease awareness, (b) sputum clearance treatments, (c) pursed lip breathing training, (d) upper-limb exercise with breathing pranayama, (e) walking training with breathing pranayama, and (f) assign a pulmonary rehabilitation program coordinator.
  Other Names: Respiratory rehabilitation
  Arms: Experimental group

SUMMARY:
The purpose of this randomized controlled trial was to evaluate the effects of a respiratory rehabilitation exercise training package on dyspnea, cough, exercise tolerance, and sputum expectoration of hospitalized elderly patients with acute exacerbation of chronic obstructive pulmonary disease (AECOPD). Using purposive sampling, 61 participants were recruited and randomly assigned to either the experimental group (n = 30) or the control group (n = 31). The experimental group participants received the respiratory rehabilitation exercise training twice a day and 10-30 minutes per session for four days. The control group participants received usual care and health education. Data were collected at baseline and at the end of the four-day intervention.

DETAILED DESCRIPTION:
The respiratory rehabilitation exercise training package included: (a) Disease awareness: The doctor explained the disease to patients and their families through the chest X-ray, (b) Sputum clearance treatments: Easily understood postural drainage cards were provided to the patients and families to assist with proper sputum clearance procedures, (c) Pursed lip breathing training: Devices were provided to the patients to ensure that the breathing exercises were completed properly, (d) Upper-limb exercise with breathing pranayama: Towels were provided to the patients to assist with upper-limb exercises properly, (e) Walking training with breathing pranayama: Legs were elevated while inhaling, and returned to the position while exhaling, and (f) Assign a pulmonary rehabilitation program coordinator: Coordinators were assigned to assist the patients in nutrition management and health education.

ELIGIBILITY:
Inclusion criteria:

1. diagnosed with moderate COPD with moderate acute exacerbation
2. over 65 years of age
3. conscious clear
4. with shortness of breath or dyspnea that was not caused by heart disease, pneumothorax, or pulmonary edema
5. had received bronchodilator aerosol therapy or antibiotic treatment, but had not been treated with an antitussive

Exclusion Criteria:

1. unstable vital signs
2. blood oxygen concentration lower than 90%
3. unstable psychological status, hemoptysis, pneumothorax, pulmonary edema, or using the respirator

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in dyspnea at 4th day | At baseline and at the 4th day of the study
  Measured by the Borg Rating of Perceived Exertion Scale.

SECONDARY OUTCOMES:
Change from baseline in cough severity at 4th day | At baseline and at the 4th day of the study
  Measured by the visual analog scale.
Change from baseline in exercise tolerance at 4th day | At baseline and at the 4th day of the study
  Measured by the 6-minute walk distance
Change from baseline in sputum expectoration at 4th day | At baseline and at the 4th day of the study
  Assessed by recording the patients' feelings regarding sputum expectoration during the previous day.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Yu Liao, MS, Principal Investigator — Chest Hospital, Ministry of Health and Welfare, Taiwan
Locations (1):
- Chest Hospital, Ministry of Health and Welfare, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Liao LY, Chen KM, Chung WS, Chien JY. Efficacy of a respiratory rehabilitation exercise training package in hospitalized elderly patients with acute exacerbation of COPD: a randomized control trial. Int J Chron Obstruct Pulmon Dis. 2015 Aug 27;10:1703-9. doi: 10.2147/COPD.S90673. eCollection 2015. PMID 26345529